CLINICAL TRIAL: NCT00876512
Title: CYP2C19 Gene Alteration and Thienopyridine Resistance in Percutaneous Coronary Intervention Study
Acronym: CALDERA-PCI
Status: Completed | Type: Observational
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Hisao Ogawa, Professor, Department of Cardiovascular Medicine, Kumamoto University
Other Study IDs: 0124
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Stable Angina
Keywords: thienopyridine resistance; stable effort angina; platelet activation; ADAMTS13; von Willebrand Factor
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CYP2C19 gene alteration is measured by using whole blood in patients with stable effort angina undergoing PCI.
Oversight: Data Monitoring Committee: No

SUMMARY:
Dual antiplatelet therapy with aspirin and thienopyridines decreases the rate of stent thrombosis in patients undergoing percutaneous coronary intervention (PCI). However, despite intensified antiplatelet treatment, some of the patients undergoing PCI develop thrombotic stent occlusion, suggesting incomplete platelet inhibition due to thienopyridine resistance. The present study is designed in order to clarify the influence of CYP2C19 genetic polymorphism on the several biomarkers for platelet activation in Japanese patients treated with thienopyridines undergoing elective PCI.

DETAILED DESCRIPTION:
We enrolled patients with stable effort angina who received dual-antiplatelet therapy with both aspirin (100mg) and clopidogrel (75mg). We performed PCI 12-24 hours after 300mg loading dose of clopidogrel, or at least 7 days of 75mg clopidogrel treatment after 300mg initial loading dose. We examined platelet adhesiveness, plasma biomarkers for platelet activation such as plasma VWF and ADAMTS13, CD40L, P-Selectin levels, and ADP-induced platelet aggregation using Light transmittance aggregometry (LTA) and VerifyNow P2Y12 assay system in those patients. We also analyzed the CYP2C19 genetic polymorphism to examine the influence of this genetic variation on the several biomarkers for platelet activation.

ELIGIBILITY:
Inclusion Criteria:

* The stable effort angina patients
* More than 20 years old
* Undergoing elective PCI treated with aspirin and clopidogrel

Exclusion Criteria:

* Patients treated with the following medical therapy (ie. Warfarin, Steroid, thrombolytic drug, Ticlopidine, Sarpogrelate hydrochloride or Cilostazol)
* Patients with the following diseases (deep vein thrombosis, atrial fibrillation, collagen disease, infection, liver or renal dysfunction, malignant diseases)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kumamoto University Hospital, Kumamoto Chuo Hospital and Saisekai Kumamoto Hospital
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Platelet function tests | before, immediately after, 1, 2, and 28 days after elective PCI
  Platelet function tests and assays for blood biomarkers of coagulation activation and inflammation before, immediately after, 1, 2, and 28 days after elective PCI.

CONTACTS AND LOCATIONS:
Locations (1):
- Kumamoto University Hospital, Kumamoto, Kumamoto, Japan